CLINICAL TRIAL: NCT02931331
Title: The Impact of Coronary Revascularization on Absolute Myocardial Blood Flow as Assessed by Stress Myocardial Positron Tomography
Brief Title: Coronary Revascularization Assessed by Stress PET
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ochsner Health System (Other)
Collaborators: Bracco Corporate (Industry)
Responsible Party: Principal Investigator, Robert Bober, M.D., Principle Investigator, Ochsner Health System
Other Study IDs: Pro00011114
Record Dates: First submitted 2016-07-06; First posted 2016-10-13 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Coronary Stenoses; Myocardial Ischemia; Coronary Artery Stenosis; Coronary Disease; Coronary Occlusion
MeSH Terms: conditions — Coronary Stenosis; Myocardial Ischemia; Coronary Disease; Coronary Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Patients undergoing standard of care (PET stress testing followed by mechanical revascularization) are undergoing an additional PET stress test to determine the impact of revascularization.

SUMMARY:
Regional absolute myocardial blood flow during stress (sMBF) as measured by Positron Emission Tomography (PET) improves post mechanical revascularization provided there is a baseline stress induced perfusion defect. Coronary revascularization performed on regions without a stress induced perfusion defect does not increase the sMBF.

DETAILED DESCRIPTION:
1.0 HYPOTHESIS Regional absolute myocardial blood flow during stress (sMBF) as measured by Positron Emission Tomography (PET) improves post mechanical revascularization provided there is a baseline stress induced perfusion defect. Coronary revascularization performed on regions without a stress induced perfusion defect does not increase the sMBF.

2.0 BACKGROUND Angiographic severity of coronary artery stenosis has historically been the primary guide to mechanical revascularization and/or medical management of coronary artery disease. Studies have shown that in patients with stable coronary artery disease (CAD) percutaneous coronary intervention (PCI) based on angiographic stenosis severity does not reduce coronary events more than initial medical treatment. In contrast, randomized trials of PCI report better outcomes when guided by fractional flow reserve (FFR) than when guided by angiographic severity or when compared to initial medical treatment.

Several potential explanations have been proposed for these conflicting views. Revascularization procedures may not alter the natural history of multicentric plaque rupture determined by complex arterial vascular biology. CAD exists diffusely in addition to segmental stenosis, so that localized mechanical intervention may fail to alter long-term disease progression or outcome. Additionally, anatomic severity on coronary angiography may not reflect the physiologic severity that directly determines ischemia, left ventricular function, and prognosis. Invasive physiologic criteria such as fractional flow reserve (FFR) can be utilized during invasive angiography to further educate decision making about whether to perform PCI, however FFR is performed in only 6% of percutaneous coronary interventions (PCI) in the United States. Consequently, percent stenosis on coronary angiography remains the main determinant when deciding to proceed with PCI.

It is well established that coronary angiography is frequently unable to adequately characterize the hemodynamic impact of coronary stenoses. In particular, percent stenosis does not predict or reliably relate to maximum flow capacity or coronary flow reserve (CFR). Studies have clearly demonstrated that the anatomical assessment of the hemodynamic significance of coronary stenoses determined by visual modalities such as coronary angiography or computed tomography coronary angiography (CTCA) does not correlate well with the functional assessment of FFR. It is plausible, therefore, that when epicardial vessels are targeted for revascularization based on percent stenosis, this intervention may not lead to a significant improvement in myocardial blood flow and in fact could be detrimental.

Myocardial perfusion by positron emission tomography (PET) is a well-established and validated tool for assessing myocardial perfusion and quantifying absolute myocardial blood flow. As such, cardiac PET serves as an ideal technology for quantifying changes in flow after revascularization procedures. Noninvasive myocardial perfusion imaging by positron emission tomography (PET) combines high spatial resolution (down to secondary or tertiary coronary branches) with quantitative measures of rest and stress myocardial perfusion in absolute units to compute absolute coronary flow reserve (CFR). Quantitative myocardial perfusion by PET has an extensive and technically robust literature, with over 250 papers including almost 15,000 subjects in the past 25 years.

Furthermore, there is robust data demonstrating prognostic information obtained from stress myocardial perfusion imaging. However, as counterintuitive and antithetical to modern practice as it seems, there are no prospective studies demonstrating that mechanical revascularization on patients with moderate or high risk perfusion scans alters prognosis. In fact, the ongoing International Study of Comparative Health Effectiveness with Medical and Invasive Approaches (ISCHEMIA) trial seeks to determine this very question. This study seeks to determine the regional effects of mechanical revascularization on patients with abnormal cardiac PET stress tests who were referred to angiography.

3.0 Study Design and Population This is a prospective, single center study from the Ochsner Medical Center. Adult patients with a stress induced perfusion defect on myocardial PET scanning who undergo mechanical revascularization will be asked to undergo a subsequent myocardial PET scan after mechanical revascularization is completed. Socio-demographic data will also be collected from the participant's electronic medical record.

4.0 Study Procedures All participants eligible for inclusion will be identified and asked to enroll with a goal of 50 participants. All Individuals will have already had an initial cardiac PET stress test (PET 1) followed by mechanical revascularization as part of their routine medical care. Enrolled participants will then be asked to perform a second cardiac PET stress test (PET 2) within 12 weeks of their revascularization procedure(s). The stress agents, radiotracer and protocol of PET 1 and PET 2 will be identical and have been described in previous studies.

5.0 Measurements Baseline absolute coronary flow and CFR will be obtained for each major coronary artery territory [left anterior descending (LAD), left circumflex (LCx), right coronary (RCA)] using FDA-approved software. Vessels will be divided into two groups: 1) those in which the baseline perfusion defect matched the revascularized territory and 2) those in which there was no baseline defect in the revascularized territory. The change in pre-vascularization and post-vascularization myocardial blood flow will be compared between the two groups. Chart review and participant interviews will include patient demographics, complete medical history, physical examination, laboratory data, 12-lead electrocardiogram (ECG), Canadian Cardiovascular Society grading of angina pectoris, and procedure reports for LHC and revascularization procedures.

6.0 Statistical Analysis Paired t-test of the average change in absolute myocardial flow between the matched and unmatched revascularized territories will be performed using SPSS software. Participant groups will be compared using Student's t-test (for normally distributed variable) or Wilcoxon's rank-sum test (for other variables) for continuous variables and the X2 test or Fisher's exact test for categorical variables. A P value of less than 0.05 will be considered statistically significant. Multiple logistic regressions will be used to determine the association between revascularization and sMBF.

7.0 Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others This study deviates from standard of care in that one additional, not clinically indicated PET stress test, will be performed soon after mechanical revascularization. Adverse events or unanticipated problems will be reported to Robert Bober, MD or Fahad Javed, MD at 504-842-2420 and the Internal Review Board as directed by Ochsner Medical Center IRB rules and regulations. Furthermore, after the first 25 patients have completed PET 2, review of adverse events and unanticipated problems will be reviewed by a safety monitoring committee comprised of 3 cardiologists who are not involved with study.

8.0 Radiation Risks Participants who enroll in the study will receive additional ionizing radiation. The effective dose of a cardiac PET scan is 5mSV or less. This is about 1/10 or 10% of the occupational exposure allowed for a radiation worker. This is also about twice the annual amount of natural background radiation exposure.

9.0 Study Withdrawal/Discontinuation Participants opting to withdraw from the study will not have the PET 2 performed.

10.0 Privacy/Confidentiality Issues All hard copies of participant data will be kept securely the PET department where only PET and research staff has access. All PET workstations are encrypted and password protected. All participant data and PET results will be de-identified of individual health information.

11.0 Follow-up and Record Retention This study is estimated to take approximately 9 months to obtain a total of 50 participants. Hard copies of PET scans are kept securely the PET department where only PET and research staff has access. The electronic PET data is encrypted and password protected. Only study personnel will have access to the files.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who undergo cardiac stress PET and subsequently undergo coronary angiography and mechanical revascularization. Mechanical revascularization is defined as PCI and/or coronary artery bypass grafting (CABG).
* Adults ≥18 and able to give informed consent.

Exclusion Criteria:

* Individuals with acute ST-elevation myocardial infarction (< 3 days)
* Individuals where absolute flow data is not available on the initial PET stress.
* Individuals who are unable to perform PET scanning secondary to hemodynamic instability.
* Individuals who are medically noncompliant with post revascularization drug therapy.
* Women who are pregnant at the time of PET2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who undergo cardiac stress PET and subsequently undergo coronary angiography and mechanical revascularization. Mechanical revascularization is defined as PCI and/or coronary artery bypass grafting (CABG).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Absolute Myocardial Flow (CC/Min/GM) | Within 12 Weeks
  Baseline absolute coronary flow and CFR will be obtained for each major coronary artery territory [left anterior descending (LAD), left circumflex (LCx), right coronary (RCA)] using FDA-approved software pre- and post-revascularization. The change in pre-vascularization and post-vascularization myocardial blood flow and relative perfusion defects will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bober, M.D., Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Medical Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boden WE, O'Rourke RA, Teo KK, Hartigan PM, Maron DJ, Kostuk WJ, Knudtson M, Dada M, Casperson P, Harris CL, Chaitman BR, Shaw L, Gosselin G, Nawaz S, Title LM, Gau G, Blaustein AS, Booth DC, Bates ER, Spertus JA, Berman DS, Mancini GB, Weintraub WS; COURAGE Trial Research Group. Optimal medical therapy with or without PCI for stable coronary disease. N Engl J Med. 2007 Apr 12;356(15):1503-16. doi: 10.1056/NEJMoa070829. Epub 2007 Mar 26. PMID 17387127
- [Background] Tonino PA, Fearon WF, De Bruyne B, Oldroyd KG, Leesar MA, Ver Lee PN, Maccarthy PA, Van't Veer M, Pijls NH. Angiographic versus functional severity of coronary artery stenoses in the FAME study fractional flow reserve versus angiography in multivessel evaluation. J Am Coll Cardiol. 2010 Jun 22;55(25):2816-21. doi: 10.1016/j.jacc.2009.11.096. PMID 20579537
- [Background] De Bruyne B, Pijls NH, Kalesan B, Barbato E, Tonino PA, Piroth Z, Jagic N, Mobius-Winkler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd KG, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Juni P, Fearon WF; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI versus medical therapy in stable coronary disease. N Engl J Med. 2012 Sep 13;367(11):991-1001. doi: 10.1056/NEJMoa1205361. Epub 2012 Aug 27. PMID 22924638
- [Background] Dattilo PB, Prasad A, Honeycutt E, Wang TY, Messenger JC. Contemporary patterns of fractional flow reserve and intravascular ultrasound use among patients undergoing percutaneous coronary intervention in the United States: insights from the National Cardiovascular Data Registry. J Am Coll Cardiol. 2012 Dec 4;60(22):2337-9. doi: 10.1016/j.jacc.2012.08.990. No abstract available. PMID 23194945
- [Background] Gould KL. Does coronary flow trump coronary anatomy? JACC Cardiovasc Imaging. 2009 Aug;2(8):1009-23. doi: 10.1016/j.jcmg.2009.06.004. PMID 19679290
- [Background] White CW, Wright CB, Doty DB, Hiratza LF, Eastham CL, Harrison DG, Marcus ML. Does visual interpretation of the coronary arteriogram predict the physiologic importance of a coronary stenosis? N Engl J Med. 1984 Mar 29;310(13):819-24. doi: 10.1056/NEJM198403293101304. PMID 6700670
- [Background] Meijboom WB, Van Mieghem CA, van Pelt N, Weustink A, Pugliese F, Mollet NR, Boersma E, Regar E, van Geuns RJ, de Jaegere PJ, Serruys PW, Krestin GP, de Feyter PJ. Comprehensive assessment of coronary artery stenoses: computed tomography coronary angiography versus conventional coronary angiography and correlation with fractional flow reserve in patients with stable angina. J Am Coll Cardiol. 2008 Aug 19;52(8):636-43. doi: 10.1016/j.jacc.2008.05.024. PMID 18702967
- [Background] Bober RM, Thompson CD, Morin DP. The effect of coronary revascularization on regional myocardial blood flow as assessed by stress positron emission tomography. J Nucl Cardiol. 2017 Jun;24(3):961-974. doi: 10.1007/s12350-016-0442-2. Epub 2016 Mar 28. PMID 27021385
- [Background] Gould KL. Positron emission tomography in coronary artery disease. Curr Opin Cardiol. 2007 Sep;22(5):422-8. doi: 10.1097/HCO.0b013e3281fc9835. PMID 17762543
- [Background] Sdringola S, Johnson NP, Kirkeeide RL, Cid E, Gould KL. Impact of unexpected factors on quantitative myocardial perfusion and coronary flow reserve in young, asymptomatic volunteers. JACC Cardiovasc Imaging. 2011 Apr;4(4):402-12. doi: 10.1016/j.jcmg.2011.02.008. PMID 21492816
- [Background] Gould KL, Johnson NP, Bateman TM, Beanlands RS, Bengel FM, Bober R, Camici PG, Cerqueira MD, Chow BJW, Di Carli MF, Dorbala S, Gewirtz H, Gropler RJ, Kaufmann PA, Knaapen P, Knuuti J, Merhige ME, Rentrop KP, Ruddy TD, Schelbert HR, Schindler TH, Schwaiger M, Sdringola S, Vitarello J, Williams KA Sr, Gordon D, Dilsizian V, Narula J. Anatomic versus physiologic assessment of coronary artery disease. Role of coronary flow reserve, fractional flow reserve, and positron emission tomography imaging in revascularization decision-making. J Am Coll Cardiol. 2013 Oct 29;62(18):1639-1653. doi: 10.1016/j.jacc.2013.07.076. Epub 2013 Aug 28. PMID 23954338
- [Background] Salerno M, Beller GA. Noninvasive assessment of myocardial perfusion. Circ Cardiovasc Imaging. 2009 Sep;2(5):412-24. doi: 10.1161/CIRCIMAGING.109.854893. No abstract available. PMID 19808630